CLINICAL TRIAL: NCT00000860
Title: Effects of Treatment for MAC Infection on Cytokine Expression in HIV-Infected Persons.
Brief Title: The Effects of Treatment for Mycobacterium Avium Complex (MAC) on the Cells of HIV-Infected Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG 853
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-07

CONDITIONS: Mycobacterium Avium-Intracellulare Infection; HIV Infections
Keywords: Tumor Necrosis Factor; AIDS-Related Opportunistic Infections; Mycobacterium avium-intracellulare Infection; Drug Therapy, Combination; Anti-HIV Agents
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; AIDS-Related Opportunistic Infections

STUDY DESIGN:
Observational Model: Natural History

SUMMARY:
To determine if treatment of MAC infection in HIV-1 infected persons is associated with the decreases in plasma levels of TNF-alpha.

Infection with MAC is a poor prognostic indicator in persons with AIDS. Evidence suggests that this poor outcome is not simply a reflection of greater immune impairment in AIDS patients with MAC infection, but rather may be a direct or indirect consequence of infection with mycobacterium. Survival of AIDS patients with MAC is shorter than those without MAC. Studies show that treatment for MAC improves the survival of MAC infected patients to nearly the survival of AIDS patients without MAC. Treatment of MAC with clarithromycin containing regimens is associated with decreased symptoms and prolonged survival. There is evidence, however, that mycobacterial infection may enhance propagation of the human immunodeficiency virus through mechanisms that may involve enhanced expression of pro inflammatory cytokines. It is unclear to what extent cytokine abnormalities contribute to this symptom complex and to what extent treatment of MAC infection will reverse these cytokine abnormalities.

DETAILED DESCRIPTION:
Infection with MAC is a poor prognostic indicator in persons with AIDS. Evidence suggests that this poor outcome is not simply a reflection of greater immune impairment in AIDS patients with MAC infection, but rather may be a direct or indirect consequence of infection with mycobacterium. Survival of AIDS patients with MAC is shorter than those without MAC. Studies show that treatment for MAC improves the survival of MAC infected patients to nearly the survival of AIDS patients without MAC. Treatment of MAC with clarithromycin containing regimens is associated with decreased symptoms and prolonged survival. There is evidence, however, that mycobacterial infection may enhance propagation of the human immunodeficiency virus through mechanisms that may involve enhanced expression of pro inflammatory cytokines. It is unclear to what extent cytokine abnormalities contribute to this symptom complex and to what extent treatment of MAC infection will reverse these cytokine abnormalities.

All patients diagnosed with MAC and who will initiate at least a 2 drug clarithromycin containing MAC treatment regimen will be eligible for participation. Blood and urine will be obtained from each patient at the following timepoints: Pre-Entry (within 7 days prior to study entry), week 4, and week 8. Sites will process and ship specific samples to Case Western Reserve University (CWRU). Various assays and analyses will be performed by CWRU. NOTE: Patients will receive no treatment on this study, however, all patients must be receiving at least a 2 drug clarithromycin containing treatment regimen for MAC either as part of participation in other studies or as prescribed by the subject's health care provider.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Patients should have successfully completed therapy or be on stable therapy for any acute infectious processes other than MAC prior to study entry.

Patients must have:

* Documented HIV infection.
* Either symptomatic MAC disease as defined by a history of clinical signs and symptoms, plus one blood culture positive for MAC or AFB obtained within the previous 90 days, OR asymptomatic MAC disease as defined by 2 blood cultures positive for MAC or AFB obtained within 90 days of entry.
* Signed parental consent for patients less than 18 years of age.

Prior Medication:

Allowed:

* Patients who have received presumptive or empiric antimycobacterial therapy prior to study entry may be enrolled if they have been treated for no more than 72 hours prior to study entry.
* Patients who have been receiving prophylaxis with azithromycin, clarithromycin and/or rifabutin may be enrolled.
* Patients should have successfully completed therapy or be on stable therapy for any acute infectious processes other than MAC prior to study entry.

Required:

* Patients must be on a stable antiretroviral regimen (same drug or combination drugs; dose modifications allowed) for at least 4 weeks prior to study entry.

NOTE:

* Patients will be requested NOT to modify or add new drugs to their stable ARV regimen for the duration of this study. Patients who absolutely require ARV changes at any time prior to week 8 will continue on study, however, their data will be analyzed separately.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Previous enrollment and permanent study drug discontinuation in ACTG 223.

Note:

* Co-enrollment in ACTG 223 and ACTG 853 is acceptable, however enrollment in both studies must be simultaneous.
* This protocol does not meet federal requirements governing prisoner participation in clinical trials and should not be considered by local IRBs for the recruitment of prisoners.

Concurrent Medication:

Excluded:

* Cytokine inhibitors.
* Corticosteroids.
* Thalidomide.
* Pentoxifylline or any other immunomodulator.
* Any interleukin.
* Colony stimulating factors (G-CSF or GM-CSF)

Patients with the following prior conditions will be excluded:

* Subjects who have had an opportunistic infection (other than MAC) within 14 days immediately preceding study entry.

Prior Medication:

Excluded within the 14 days immediately preceding study entry:

* Cytokine inhibitors.
* Corticosteroids.
* Thalidomide.
* Pentoxifylline or any other immunomodulator.
* Any interleukin.
* Colony stimulating factors (G-CSF or GM-CSF)

Prior Treatment:

Excluded:

* Patients who have received a blood transfusion within the 14 days immediately preceding study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24

CONTACTS AND LOCATIONS:
Overall Officials: MacArthur R, Study Chair; Benson C, Study Chair; Lederman M, Study Chair
Locations (11):
- United States (11):
  - San Francisco Gen Hosp, San Francisco, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Washington Reg AIDS Prog / Dept of Infect Dis, Washington D.C., District of Columbia
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Univ of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Benson CA. MAC: pathogenesis and treatment. Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:166
- [Background] MacArthur RD, Lederman MM, Benson CA, Chernoff MC, MacGregor RR, Spritzler J, Mahon LF, Yen-Lieberman B, Purvis S. Effects of Mycobacterium avium complex-infection treatment on cytokine expression in human immunodeficiency virus-infected persons: results of AIDS clinical trials group protocol 853. J Infect Dis. 2000 Apr;181(4):1486-90. doi: 10.1086/315370. Epub 2000 Apr 13. PMID 10762582
- [Background] MacArthur RD, Lederman M, Benson CA, Chernoff MC, Mahon LF, Yen-Lieberman B, Purvis S, MacGregor RR. ACTG 853: effects of treatment for MAC infection on cytokine expression in HIV-infected persons. Intersci Conf Antimicrob Agents Chemother. 1998 Sep 24-27;38:403 (abstract no I-130)